CLINICAL TRIAL: NCT01889329
Title: Development and Field Testing of Ready-to-use-therapeutic Foods Made of Local Ingredients in Bangladesh for the Treatment of Children With Severe Acute Malnutrition
Brief Title: Development and Field Testing of Ready-to-use-therapeutic Foods Made of Local Ingredients in Bangladesh for SAM Children
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: UNICEF (Other); Nutriset (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PR-11005
Record Dates: First submitted 2013-06-26; First posted 2013-06-28 (Estimated); Last update posted 2022-02-11 (Actual); Status verified 2015-06

CONDITIONS: Severe Acute Malnutrition in Childhood

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- RUTF-1 (Experimental): Made from local food ingredients
  Interventions: Dietary Supplement: RUTF-1
- RUTF-2 (Experimental): Made from local food ingredients
  Interventions: Dietary Supplement: RUTF-2
- Plumpynut (Active Comparator): Made from peanut
  Interventions: Dietary Supplement: Plumpynut

INTERVENTIONS:
Dietary Supplement: RUTF-1 — Made from local food ingredients
  Arms: RUTF-1
Dietary Supplement: RUTF-2 — Made from local food ingredients
  Arms: RUTF-2
Dietary Supplement: Plumpynut — Commercially made from peanut paste
  Arms: Plumpynut

SUMMARY:
Around 0.5 million under-five children are currently suffering from severe acute malnutrition (SAM) in Bangladesh and are at risk of death. Children with SAM and complications should be treated in a health care facility. It is imperative, however, to manage children with SAM but without any complications in the community. This requires a ready-to-use-therapeutic food (RUTF) that conforms to standard recommendations on its composition. The prototype RUTF is peanut based, made outside Bangladesh, and has to be imported. By developing a RUTF using local food ingredients, test it for acceptability and efficacy in the treatment of children with SAM, hopefully make the treatment of SAM cost-effective and sustainable.

Hypothesis: Does the locally developed ready-to-use-therapeutic foods (RUTFs) demonstrate similar or better acceptability and efficacy in the treatment of children suffering from severe acute malnutrition (SAM) when compared to the prototype RUTF (Plumpynut)?

DETAILED DESCRIPTION:
Childhood malnutrition continues to be a significant public health problem in the world, especially in Asia. Acute malnutrition and more so, severe acute malnutrition (SAM) among children below five years of age remains a major embarrassment, and impediment to optimal human capital development in Asia. Without access to appropriate treatment, these SAM children are at high risk of death; there are only a few hospitals in Bangladesh and other developing countries with facilities for managing these children appropriately and their coverage is extremely low. In 2008, the Government of Bangladesh published National Guidelines for management of SAM at the facility level. However, these national guidelines have yet to become operationalized and there are very small exploratory initiatives that focus on community-based management of acute malnutrition (CMAM). Under the auspices of the Directorate General of Health Services, a 2007 national consensus meeting on the management of SAM resolved that CMAM along with scaling up facility-based management is essential for Bangladesh but that a local RUTF should be developed to ensure cost-effective and sustainable programs. Absence of a RUTF that is made of locally available food ingredients and hence, relatively inexpensive, is impeding the implementation of programs for community-based management of SAM in the country. The proposed project will develop new and improved recipes of RUTF based on established principles of dietetics and select at least two candidate RUTFs for treating SAM and testing their acceptability and efficacy. The experiments for development of RUTF will be done in ICDDR,B Food Processing Laboratory by the investigators. Experiments, including assessment of the composition of the local food ingredients and the presence of anti-nutrient factors, such as phytate, will be performed in the laboratories of Nutriset in France. Acceptability of the candidate RUTFs by the children as well as by the mothers will be assessed and compared among groups of children, who receive any new two RUTF products and the prototype RUTF (Plumpy'nut). For efficacy trial, the study population will be the children who will come to ICDDR,B hospital with SAM and complications. They will receive the standardized management during the acute/initial phase of treatment in the hospital. After completion of the initial treatment of associated medical complications an appetite test with the standard RUTF will be done. If the child passes the appetite test, the child will be enrolled in the study and subsequent alternate feeds of the child will be replaced with the assigned RUTF. The child will be further observed next day giving the total ration of the assigned RUTF and will be monitored for any possible adverse effects, e.g. skin rash, urticaria from food allergy, abdominal distension, pain abdomen, vomiting, diarrhea or any other significant change in clinical status. If there is no unwanted event and the child eats RUTF eagerly, then the child will be discharged from the hospital with RUTF ration for one week (7- 10 days' ration covering the weekends and any holidays). The RUTFs will be used in a partial double-blind manner. Complete blinding of the three RUTFs might not be possible because of distinctive smell of peanuts in proto type RUTF. Other two candidate RUTFs will be blinded. The code will be kept by the producer of the sachets (Nutriset) and Dr ASG Faruque, Senior Scientist, ICDDR'B, who will not be involved with the study. A team of ICDDR,B staff will be responsible for implementation of the study. All field personnel recruited will be full time for this study and will have prior experience in interview techniques, data collection, and assessment of nutritional status. Before starting field activities, an intensive 5-day training will be given to the supervisors and interviewers. The quality control team supported by investigator(s) will monitor the performance of field personnel through regular observation at the household level and regular checks of data for completeness. The quality control team will independently check the data collection. Errors detected will be corrected immediately in the field. The entire assignment including the report writing will be completed within 24 months after the IRB approval from ICDDR,B and signing of MOU between the UNICEF, Bangladesh, Nutriset and ICDDR,B.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 to 59 months (either sex)
* Suffering from Severe Acute Malnutrition (SAM) defined by WHZ <-3 using WHO growth standards 2006 and/or having bipedal edema (nutritional), and/or MUAC <11.5 cm
* Have completed acute (stabilization) phase management, are clinically well, and have an appetite
* Additional enrollment criteria will be: no signs of concurrent infection, mothers/caregivers agree to stay in their current address for at least the next three months (for ease of follow-up of the children)
* Informed written consent obtained from the parent or guardian.

Exclusion Criteria:

* Failure to obtain Informed consent from parents or caretakers
* Children without any fixed address
* Children with tuberculosis (diagnosis based on WHO 2006 guidelines which have been incorporated in the national TB control guidelines of Bangladesh)
* Any congenital/acquired disorder affecting growth i.e. trisomy-21 or cerebral palsy
* Children on an exclusion diet for the treatment of persistent diarrhea
* Having known history of soy, peanut or milk protein allergy.

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 490 (Actual)
Dates: Start 2013-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Weight gain (g/kg/d) | Initially 3 months for the acceptability trial another 18 months will be required for the efficacy trial
  The primary objective of the proposed study will be to develop ready-to-use therapeutic food (RUTF) that will ultimately be used to treat childhood severe acute malnutrition which continues to be highly prevalent in Bangladesh. This will involve selection of candidate recipes of RUTF and testing them for acceptability and efficacy among children and caregivers. The successful candidate recipe of local RUTF is expected to have better weight gain (g/kg/d) in children suffering from Severe Acute Malnutrition (SAM).

CONTACTS AND LOCATIONS:
Locations (1):
- International Centre for Diarrhoeal Disease Research, Bangladesh (icddr,b), Dhaka, Bangladesh

REFERENCES:
- [Derived] Weagley JS, Zaydman M, Venkatesh S, Sasaki Y, Damaraju N, Yenkin A, Buchser W, Rodionov DA, Osterman A, Ahmed T, Barratt MJ, DiAntonio A, Milbrandt J, Gordon JI. Products of gut microbial Toll/interleukin-1 receptor domain NADase activities in gnotobiotic mice and Bangladeshi children with malnutrition. Cell Rep. 2022 Apr 26;39(4):110738. doi: 10.1016/j.celrep.2022.110738. PMID 35476981